CLINICAL TRIAL: NCT02130726
Title: The STOMACH Trial: Surgical Technique, Open Versus Minimally-invasive Gastrectomy After CHemotherapy
Brief Title: Surgical Technique, Open Versus Minimally-invasive Gastrectomy After CHemotherapy
Acronym: STOMACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Stichting Nuts Ohra (Other)
Responsible Party: Principal Investigator, J. Straatman, MD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STOMACH trial
Record Dates: First submitted 2014-04-28; First posted 2014-05-05 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Minimally-invasive; Oncological quality of resection
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minimally-invasive Gastrectomy (Experimental): Patients allocated to the 'Minimally-invasive Gastrectomy' group will undergo minimally-invasive/laparoscopic total gastrectomy. If, during surgery, laparoscopic resection does not seem feasible, the procedure may be converted to an open one.
  Interventions: Procedure: Minimally-invasive gastrectomy
- Open Gastrectomy (Active Comparator): Patients allocated to the 'Open Gastrectomy' group will receive total resection of the stomach via laparotomy. This group is considered the control group
  Interventions: Procedure: Open Gastrectomy

INTERVENTIONS:
Procedure: Minimally-invasive gastrectomy — Patients allocated to the 'Minimally-invasive gastrectomy' arm will receive total gastrectomy via laparoscopy.
  Other Names: laparoscopic gastrectomy
  Arms: Minimally-invasive Gastrectomy
Procedure: Open Gastrectomy — patients allocated to the 'Open gastrectomy' group will receive total gastrectomy via laparotomy
  Other Names: Conventional Gastrectomy
  Arms: Open Gastrectomy

SUMMARY:
Laparoscopic surgery has been shown to provide important advantages in comparison with open procedures in the treatment of several malignant diseases, such as less peri-operative blood loss, faster patient recovery and shorter hospital stay. All while maintaining similar results with regard to tumour resection margin and oncological survival. In gastric cancer the role of laparoscopic surgery remains unclear.

Current recommended treatment for gastric cancer consists of radical resection of the stomach, combined with lymfadenectomy. The extent of lymfadenectomy is considered a marker for radicality of surgery and quality of care. Therefore, It is imperative that a new surgical technique should be non-inferior with regard to radicality and lymph node yield.

Preliminary studies show promising results for laparoscopic gastrectomy, but the number of studies is small and due to lower incidence of gastric cancer in the West they are often underpowered. A prospective randomised clinical trial is indicated in order to establish the optimal surgical technique in gastric cancer: open versus minimally invasive gastrectomy.

Results of the STOMACH trial will further aid in determining the optimal surgical technique in patients with gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or above 18 years
* Primary adenocarcinoma of stomach, indication for total gastrectomy with curative intent.
* Neoadjuvant therapy (epirubicin, cisplatin, capecitabine)
* Surgical resectable (T1-3, N0-1, M0)
* Informed consent

Exclusion Criteria:

* Previous or coexisting cancer
* Previous surgery of the stomach
* ASA classification (American Society of Anaesthesiologists) score 4 or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-12; Primary Completion 2019-03 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Extent of lymph node dissection | two weeks
  The extent of lymph node dissection in treatment of gastric cancer is considered a prognostic marker for postoperative survival and disease-free survival. Before implementation of a new surgical technique, it is imperative that this technique is non-inferior with regard to the extent of lymph node dissection. Measures will include the number of resected lymph nodes and the number of resected lymph node stations.

SECONDARY OUTCOMES:
Postoperative complications | Postoperatively with follow-up to one year
  Postoperative complications after major abdominal surgery, such as gastric resection, lead to increased morbidity and mortality. A new surgical technique should be non-inferior or even improve outcomes with regard to postoperative complications. Complications will be graded according to the Clavien-Dindo classification, which grades complications with regard to necessary treatment for this complication. Also Long-term complications, such as hernia cicatricialis will be monitored.
Quality of Life | 1 and 5 days postoperatively, 3 months, 6 months and 12 months
  Patient Related Outcome Measures (PROMs) are of increasing importance. A new surgical technique should aim at improved PROMs, which will be measured with several questionnaires. The SF-36 and GIQLI questionnaires.
Duration of hospital admission | during admission, average 2 weeks
  Minimally-invasive surgery is associated with faster patient recovery and shorter duration of hospital admission. The number of days of hospital admission will be recorded. Readmission will be registered separately.
Duration of Intensive Care admission | During submission, average 2 days
  Minimally-invasive surgery is associated with faster patient recovery, therefore we expect the number of days spent on the intensive care unit to be less in this group.
Peri-operative blood loss | during surgery, 1 day
  Minimally-invasive surgery is associated with less peri-operative blood loss. Blood loss will be measured in milliliters and average blood loss will be compared to the conventional 'open' group.
Duration of Surgery | Peri-operatively, 1 day
  Due to the techniques associated with minimally-invasive surgery the average procedure takes longer to complete. The duration of the procedure will be registered in minutes.
Cost-effectiveness | from surgery to one year follow-up
  Cost-effectiveness will be measured based on duration and equipment necessary for surgery, admission duration, ICU admission and reinterventions.
Disease-free survival | up to 5 years postoperatively
  In order to further assess oncological feasibility of minimally-invasive gastrectomy disease-free survival will be monitored up to 5 years postoperatively. Patients are informed, when they enter the study, that they can be contacted for additional information up to 5 years postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: D.L. van der Peet, MD, PhD, Principal Investigator — VU Medisch Centrum
Locations (8):
- Universitätsklinikum Carl Gustav Carus, Dresden, Germany
- Netherlands (2):
  - VU Medical Center, Amsterdam, NLNH
  - Academic Medical Centre, Amsterdam, North Holland
- Spain (4):
  - Hospital universitari Basurto, Bilbao
  - Hospital Jerez de la Frontera, Cadiz
  - Hospital Universitario de Josep Trueta, Girona
  - Hospital Universitario del Sureste de Madrid, Madrid
- Salford Royal NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Derived] van der Wielen N, Daams F, Rosati R, Parise P, Weitz J, Reissfelder C, Del Val ID, Loureiro C, Parada-Gonzalez P, Pintos-Martinez E, Vallejo FM, Achirica CM, Sanchez-Pernaute A, Campos AR, Bonavina L, Asti ELG, Poza AA, Gilsanz C, Nilsson M, Lindblad M, Gisbertz SS, van Berge Henegouwen MI, Romario UF, De Pascale S, Akhtar K, Cuesta MA, van der Peet DL, Straatman J. Three-year survival and distribution of lymph node metastases in gastric cancer following neoadjuvant chemotherapy: results from a European randomized clinical trial. Surg Endosc. 2023 Sep;37(9):7317-7324. doi: 10.1007/s00464-023-10278-5. Epub 2023 Jul 19. PMID 37468751
- [Derived] Straatman J, van der Wielen N, Cuesta MA, Gisbertz SS, Hartemink KJ, Alonso Poza A, Weitz J, Mateo Vallejo F, Ahktar K, Diez Del Val I, Roig Garcia J, van der Peet DL. Surgical techniques, open versus minimally invasive gastrectomy after chemotherapy (STOMACH trial): study protocol for a randomized controlled trial. Trials. 2015 Mar 27;16:123. doi: 10.1186/s13063-015-0638-9. PMID 25873249